CLINICAL TRIAL: NCT00830297
Title: Treat-to-target Trial of Basal Insulin in Post-transplant Hyperglycemia (TIP): Efficacy and Safety of a Novel Protocol in Renal Transplant Recipients Receiving a Tacrolimus-based Immunosuppression
Brief Title: Treat-to-target Trial of Basal Insulin in Post-transplant Hyperglycemia
Acronym: TIP
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Marcus Saemann (Other)
Responsible Party: Sponsor-Investigator, Marcus Saemann, Ass. Prof. Dr. Marcus Säemann, Medical University of Vienna
Organization: Medical University of Vienna (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EudraCT: 2008-005951-84
Record Dates: First submitted 2009-01-26; First posted 2009-01-27 (Estimated); Last update posted 2012-09-03 (Estimated); Status verified 2012-08

CONDITIONS: Hyperglycemia
Keywords: TIP; NODAT; hyperglycemia; long-acting insulin; post-transplant hyperglycemia
MeSH Terms: conditions — Hyperglycemia | interventions — Isophane Insulin, Human; Insulin, Long-Acting; Congresses as Topic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 Insulatard (long-acting insulin) (Active Comparator)
  Interventions: Drug: Insulatard (long-acting insulin)
- 2 Conventional treatment (Active Comparator)
  Interventions: Drug: Conventional

INTERVENTIONS:
Drug: Insulatard (long-acting insulin) — In group No.1 (study arm 1 (=A)), patients will be treated with long-acting insulin (Insulatard) as soon as the glucose-level before supper surpasses 140 mg/dl. The normoglycemic goal in this group will be from 110 to 120 mg/dl.
  Arms: 1 Insulatard (long-acting insulin)
Drug: Conventional — In group No.2 (study arm 2 (=B)), patients will be treated conventionally according to the decisions taken by the physicians on the ward. The following suggestions will be brought to the attention of the ward in order to standardize the treatment of the patients in study arm B: 1. Treatment in this group should be initiated if the fasting glucose level surpasses the renal glucose threshold, i.e. 180 mg/dl. 2. As the proposed life-style modifications for the treatment of NODAT1 are not feasible during this very early post-transplant phase, the basis of the conventional therapy will be proposed to be sulfonyl urea drugs (i.e. Gliclazide - Diamicron®, 30 mg, not more than twice daily). 3. Short-acting insulin will be strongly recommended to be used for corrections of capillary blood glucose levels above 250 mg/dl.
  Arms: 2 Conventional treatment

SUMMARY:
Treat-to-target trial of basal Insulin in Post-transplant hyperglycemia (TIP): efficacy and safety of a novel protocol in renal transplant recipients receiving a tacrolimus-based immunosuppression

DESCRIPTION:

A prospective, randomized safety and efficacy study of long-acting insulin (Insulatard®) as therapy against post-transplant hyperglycemia in renal transplant recipients

OBJECTIVES:

Primary Objective:

To demonstrate superiority of long-acting insulin (Insulatard®) against post-transplant hyperglycemia, in comparison to conventional treatment, and as evaluated by HbA1c

Secondary Objectives:

* To assess the average post-transplant glucose levels in renal transplant patients under conventional blood-glucose lowering therapy during a period of at least 14 days after transplantation by measuring the capillary blood glucose levels four times daily in both groups of patients (fasting, before lunch, before supper, after supper)
* To detect the number of post-transplant patients who - without any history of pre-transplant diabetes - develop at least one episode of post-transplant hyperglycemia (> 140 mg/dl before supper)
* To detect the average number of hyperglycemic episodes in post-transplant patients with at least one episode of post-transplant hyperglycemia and without any history of diabetes
* To assess the amount of (long-acting) insulin (in IU) needed in order to obtain a target capillary blood glucose level in the range of 110 mg/dl to 120 mg/dl before supper in post-transplant patients with incidence of hyperglycemia
* To assess the safety of long-acting insulin in controlling post-transplant hyperglycemia (especially with regards to episodes of hypoglycemia (glucose-level < 60 mg/dl)
* To assess the prevalence of post-transplant diabetes, as diagnosed by an abnormal oral glucose tolerance on days 90, 180 and 360 after transplantation, in the group of patients which has been treated with long-acting insulin, in comparison to patients who received conventional treatment
* To assess the morbidity (hospitalization, infections, subsequent episodes of surgery, requirement of non-immunosuppressive, non- blood glucose lowering medication) in the group of patients with long-acting insulin for hyperglycemia, in comparison to patients randomized into the group receiving conventional treatment
* To assess the renal outcome (creatinine levels, rejections) in the group of patients which is foreseen to be treated with long-acting insulin for hyperglycemia, in comparison to patients randomized into the group receiving conventional treatment

DETAILED DESCRIPTION:
DESIGN / PHASE:

Prospective, single-center, randomized, parallel group, controlled, phase II study.

STUDY PLANNED DURATION:

First patient First visit 1Q 2009 Last patient First visit 4Q 2009 Last patient Last visit 4Q 2010

CENTERS:

Department of Internal Medicine III, Division of Nephrology and Dialysis, Medical University of Vienna, Austria, Department of Surgery, Division of Transplantation, Medical University of Vienna, Austria

PATIENTS / GROUPS:

50 patients in 2 groups 25 patients per group Randomization ratio 1:1, no stratification

Capillary blood glucose will be measured four times daily: before breakfast (7:30 am), before lunch (12 pm), before supper (5:30 pm) and after supper (9 pm) in both groups by the nursing personnel/academic investigators. In group No.1 (study arm A), patients will be treated with long-acting insulin (Insulatard) as soon as the glucose-level before supper surpasses 140 mg/dl. The normoglycemic goal in this group will be from 110 to 120 mg/dl.

In group No.2 (study arm B), the glucose levels will be recorded, but the treatment will be left up to the ward, which is relying on conventional morning glucose measurements. For safety, any glucose levels >180 mg/dl will be reported, and all measures taken by the ward will be recorded. As there are no available guidelines however concerning the so called "conventional" blood glucose-lowering therapy in renal transplant patients, especially during this very early post-transplant phase, the following suggestions will be brought to the attention of the ward in order to standardize the treatment of the patients in study arm B: 1. Treatment in this group should be initiated if the fasting glucose level surpasses the renal glucose threshold, i.e. 180 mg/dl. 2. As the proposed life-style modifications for the treatment of NODAT1 are not feasible during this very early post-transplant phase, the basis of the conventional therapy will be proposed to be sulfonyl urea drugs (i.e. Gliclazide - Diamicron®, 30 mg, not more than three times daily). 3. Short-acting insulin will be strongly recommended to be used for corrections of capillary blood glucose levels above 250 mg/dl.

EFFICACY ENDPOINTS:

Primary:

- HbA1c levels

Secondary:

* capillary blood glucose profile in patients treated with long-acting insulin and in the control group, as evaluated by the daily measurements
* number of patients and overall number of days with hyperglycemia > 140 mg/dl (in each group)
* number of patients and overall number of days with hyperglycemia > 200 mg/dl (in each group)
* number of patients and overall number of days with hypoglycemia < 60 mg/dl in each group
* number of patients with abnormal glucose tolerance on days 90, 180 and 360 after transplantation

TOLERABILITY / SAFETY ENDPOINTS:

- Number of incidences of symptomatic hypoglycemia, confirmed by capillary blood glucose levels < 60 mg/dl

PHARMACOKINETIC / PHARMACODYNAMIC ENDPOINTS:

Doses of (long-acting) insulin

STATISTICAL METHODOLOGY:

Primary Endpoint:

HbA1c (rel %)

Null and alternative hypotheses:

H0 Treatment of hyperglycemia > 140 mg/dl before supper with long-acting insulin in renal transplant recipients for a period of at least 14 days after transplantation is equal to conventional treatment in reducing the HbA1c (measured on day 90 after transplantation).

H1: Treatment of hyperglycemia > 140 mg/dl before supper with long-acting insulin in renal transplant recipients for a period of at least 14 days after transplantation is superior to conventional treatment in reducing the HbA1c (measured on day 90 after transplantation).

Type-I and -II errors - power:

α=0.05 ß=0.2

Statistical methodology:

One-sided t-test of HbA1c on day 90 after transplantation, one-sided t-test of number of days with hyperglycemia > 140 mg/dl before supper, comparison of capillary blood glucose levels by ANOVA

Sample size calculation:

Based on a two-sided testing and an expected standard deviation of HbA1c of 10%, an α=0.05 and a ß=0.2, a sample size of 25 patients per group was determined.

Main analysis set:

Per-protocol (efficacy) and intention to treat (ITT) for safety

Other endpoints:

descriptive statistics

ELIGIBILITY:
Inclusion Criteria:

* renal transplantation (deceased or living donor)
* eligibility for the standard immunosuppression of our center, consisting of tacrolimus, mycophenolate mofetil or mycophenolic acid, dexamethasone/prednisone triple therapy
* informed consent of the patient

Exclusion Criteria:

* patients with type 1 or type 2 diabetes
* allergy against long-acting insulin

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2009-01; Primary Completion 2010-12 (Actual); Study Completion 2011-05 (Actual)

PRIMARY OUTCOMES:
The primary endpoint is the difference in HbA1c between the two study arms. | post-transplant day 90

SECONDARY OUTCOMES:
Capillary blood glucose profiles in each group | post-transplant day 1-21
Number of patients and overall number of days with hyperglycemia >140 mg/dl before supper (in each group) | post-transplant day 1 - 21
Number of patients and overall number of days with hyperglycemia >200 mg/dl (in each group) | post-transplant day 1-21
Number of patients and overall number of days with hypoglycemia <60 mg/dl in each group | post-transplant day 1-21
Number of patients with abnormal glucose tolerance | post-transplant day 90, 180 and 360
Difference in HbA1c between the two study arms | post-transplant day 180 and 360

CONTACTS AND LOCATIONS:
Overall Officials: Wilfred Druml, MD, Study Chair — Medical University of Vienna
Locations (1):
- Medical University of Vienna, Department of Internal Medicine III, Vienna, Austria

REFERENCES:
- [Background] Davidson JA, Wilkinson A; International Expert Panel on New-Onset Diabetes after Transplantation. New-Onset Diabetes After Transplantation 2003 International Consensus Guidelines: an endocrinologist's view. Diabetes Care. 2004 Mar;27(3):805-12. doi: 10.2337/diacare.27.3.805. No abstract available. PMID 14988309
- [Derived] Lo C, Toyama T, Oshima M, Jun M, Chin KL, Hawley CM, Zoungas S. Glucose-lowering agents for treating pre-existing and new-onset diabetes in kidney transplant recipients. Cochrane Database Syst Rev. 2020 Jul 30;8(8):CD009966. doi: 10.1002/14651858.CD009966.pub3. PMID 32803882